CLINICAL TRIAL: NCT04126135
Title: Comparative Effectiveness of Cystine Versus Nicotine Replacement Therapy (NRT) in the National Smoking Cessation Program of Mongolia: A Pragmatic Non-Inferiority Trial
Brief Title: Comparative Effectiveness of Cystine Versus Nicotine Replacement Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Pfizer (Industry); Mongolian National University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pramil N Singh, Director and Professor, Transdisciplinary Tobacco Research Program, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5170400
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nicotine Addiction
Keywords: Smoking Cessation, Nicotine Replacement Therapy, Cytisine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — cytisine; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Group (Active Comparator): Subjects are asked to completely stop smoking on their quit day and use a daily Nicotine Replacement Therapy (NRT) patch for 25 days.
  Interventions: Drug: Nicotine Replacement Therapy (NRT)
- Treatment Group (Experimental): Subjects will start a 25-day course of Cytisine tablets started during the four days before the quit date and are asked to reduce smoking during this time.
  Interventions: Drug: Cytisine

INTERVENTIONS:
Drug: Cytisine — Subjects will take a 25-day course of Cytisine tablets started during the 4 days before the quit date. They will be asked to reduce smoking during this time.
  Arms: Treatment Group
Drug: Nicotine Replacement Therapy (NRT) — Subjects are asked to completely stop smoking on their quit day and use a daily NRT patch for 25 days.
  Arms: Usual Care Group

SUMMARY:
A pragmatic, single blinded, randomized, controlled non-inferiority trial of Cytisine versus Nicotine Replacement Therapy for continuous abstinence is conducted in the government run primary health hospitals in Mongolia.

DETAILED DESCRIPTION:
Rationale: In Mongolia, smoking cessation assistance in the governmental health sector consists of behavioral counseling and a 3-week regimen of the NRT patch that costs 175 USD. This cost for low income adults limits effectiveness. A 2014 study documented the superiority and lower cost (<20 USD) of Cytisine versus NRT for continuous abstinence. Trial investigators are testing the comparative effectiveness of Cytisine in the "real life setting" of their national health care system and, if proven effective, will include coverage for Cytisine in the national health plan.

Research Question/Objective: To determine whether a 25 day course of Cytisine tablets is at least as effective as 25 days of NRT in helping smokers remain abstinent for at least one month.

Design: A pragmatic, single blinded, randomized, controlled non-inferiority trial.

Setting: Six governmental primary care centers in Ulaanbaatar, Mongolia, and outskirts.

Participants: Mongolian adult smokers referred to government-run addiction units.

Intervention and procedures: Participants are randomized to 5 weeks of treatment (n=654) or usual care (n=653) and a 6-month follow-up. The treatment consists of a 25-day course of Cytisine tablets and behavioral counseling. Usual care consists of 25 days of NRT and behavioral counseling.

Measurements: The primary outcome is continuous abstinence (< 5 cigarettes smoked since quit date) at 1 month. Secondary outcomes include 7-day point prevalence abstinence rates and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Seeking smoking cessation treatment
* Ages 18 years or older
* Currently smoking > 5 cigarettes per day
* Willingness to make quit attempt with pharmacotherapy
* Able to provide verbal and written informed consent
* Have telephone access

Exclusion Criteria:

* Pregnancy or currently breastfeeding
* Current users of NRT (patch, gum, lozenge)
* Current users of non_NRT smoking cessation pharmacotherapy
* Enrolled in another smoking cessation program (non-governmental)
* Clinical disorder that contraindicates use of NRT or Cytisine (heart attack, stroke, severe angina within the past 2 weeks, uncontrolled hypertension, phaeochromocytoma, severe mental illness)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1307 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Length of abstinence after 25 day course of Cytisine. | One month after quit date
  Continuous abstinence is defined as <5 cigarettes smoked since quit date. Subjects will complete survey to determine number of cigarettes smoked since quit day.

SECONDARY OUTCOMES:
Length of abstinence after 25 days of NRT | One month after quit date
  Continuous abstinence is defined as <5 cigarettes smoked since quit date. Subjects will complete survey to determine number of cigarettes smoked since quit day.

CONTACTS AND LOCATIONS:
Overall Officials: Pramil N Singh, DrPH, Principal Investigator — Loma Linda University Health; Davaalkham Dambadarjaa, MD, Principal Investigator — Mongolian National University of Medical Sciences
Locations (1):
- Mongolian National University of Medical Sciences, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No